CLINICAL TRIAL: NCT03058406
Title: Special Use Investigation of HALAVEN (HAL03T) - Study on Safety and Efficacy in Patients With Soft Tissue Sarcomas
Brief Title: A Study on Safety and Efficacy in Patients With Soft Tissue Sarcomas
Acronym: HAL03T
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E7389-M081-503
Record Dates: First submitted 2017-02-16; First posted 2017-02-20 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2018-08

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Sarcoma, Soft Tissue; Halaven Injection; E7389
MeSH Terms: conditions — Sarcoma | interventions — eribulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eribulin mesylate
  Interventions: Drug: Eribulin mesylate

INTERVENTIONS:
Drug: Eribulin mesylate — Participants will receive 1.4 milligrams per square meter (mg/m2) administered as an intravenous (IV) infusion (over 2 to 5 minutes) on Days 1 and 8 of each 3-week cycle and beyond.
  Other Names: Halaven Injection; E7389

SUMMARY:
The purpose of this study is to understand safety and efficacy in participants with soft tissue sarcomas.

ELIGIBILITY:
Inclusion Criteria:

- Participants with soft tissue sarcoma who will receive eribulin mesylate per the approved indication in routine clinical practice

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with soft tissue sarcoma who will receive eribulin mesylate per the approved indication in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-11-04 (Actual); Study Completion 2018-11-04 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) and Adverse Drug Reactions (ADRs) | up to 2 years

SECONDARY OUTCOMES:
Survival Rate at Year 2 | up to 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

REFERENCES:
- [Derived] Kawai A, Narahara H, Takahashi S, Nakamura T, Kobayashi H, Megumi Y, Matsuoka T, Kobayashi E. Safety and effectiveness of eribulin in Japanese patients with soft tissue sarcoma including rare subtypes: a post-marketing observational study. BMC Cancer. 2022 May 11;22(1):528. doi: 10.1186/s12885-022-09527-y. PMID 35546669
- [Derived] Kobayashi E, Naito Y, Asano N, Maejima A, Endo M, Takahashi S, Megumi Y, Kawai A. Interim results of a real-world observational study of eribulin in soft tissue sarcoma including rare subtypes. Jpn J Clin Oncol. 2019 Oct 1;49(10):938-946. doi: 10.1093/jjco/hyz096. PMID 31365116